CLINICAL TRIAL: NCT05678153
Title: Effect of Passive Smoking on Orofacial Dysfunction Among a Group of Egyptian Children: A Cohort Study
Acronym: ACU222
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf A.Elsabour, Primary investigator, Ahram Canadian University
Other Study IDs: ACU 222
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Smoking; Orofacial Dysfunction
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- passive smokers children group (study group): children whose parents reported having one or more family members smokes indoors in the presence of the child
  Interventions: Diagnostic Test: Nordic Orofacial Test-Screen (NOT-S)
- non-passive smokers children group (control group): children whose parents reported not to have one or more family members smokes indoors in the presence of the child
  Interventions: Diagnostic Test: Nordic Orofacial Test-Screen (NOT-S)

INTERVENTIONS:
Diagnostic Test: Nordic Orofacial Test-Screen (NOT-S) — screening tool to detect orofacial dysfunction

SUMMARY:
This study aims to investigate the orofacial dysfunction in children who are subjected to passive smoking and to correlate its results to their saliva cotinine levels

DETAILED DESCRIPTION:
The participants will be recruited from the pedodontics outpatient clinic in the, Faculty of Oral and Dental Medicine, Ahram Canadian University, Egypt. The aim and the steps of the study will be explained to the guardian.

After obtaining the informed consent, the investigator will fill an administrative questionnaire, which includes parents and child's personal data, medical and dental history, a question inquiring if one of the parents smokes in the house, the frequency of smoking, smoking type, and number of cigarettes (if present).

Then, the examination of orofacial dysfunction will be evaluated by the investigator, using Nordic Orofacial Test - screen (NOT-S)

ELIGIBILITY:
Inclusion Criteria:

* Children who are free from any systematic disease, or genetic disorders that
* Children whose families accept to participate in this study.

Exclusion Criteria:

* Children whose parents quit smoking after the child was born.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cooperative Egyptian children aged from (four to seven) years.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Orofacial Dysfunction (measured using Nordic Orofacial Test-Screen) | baseline record
  deviation from normal functions of facial and oral structures

CONTACTS AND LOCATIONS:
Overall Officials: Mennat Allah Abd-Elsabour, Master, Principal Investigator — Ahram Canadian University

IPD SHARING:
Plan to Share IPD: Undecided